CLINICAL TRIAL: NCT03219411
Title: A Multi-National, Double-Blind, Randomized Trial Of The Influence Of Cinnamon Powders In Subjects With Risk For Developing Diabetes
Brief Title: Effects of Cinnamon Supplementation on Glucose Metabolism in Patients With Pre-diabetes
Acronym: Cinnamon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Kyunghee University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHS #:2017-15
Record Dates: First submitted 2017-07-11; First posted 2017-07-17 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Dysglycemia; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinnamon (Active Comparator): Cinnamon burmannii administered orally as 500-mg capsules three times daily over 12 weeks
  Interventions: Dietary Supplement: Cinnamon
- Placebo (Placebo Comparator): Placebo administered orally as capsules three times daily over 12 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Cinnamon — Cinnamon burmannii administered orally as 500-mg capsules three times a day over 12 weeks
  Arms: Cinnamon
Other: placebo — Placebo administered orally as capsules three times a day over 12 weeks
  Arms: Placebo

SUMMARY:
The transition from normal glucose tolerance to overt type 2 diabetes mellitus (T2D) encompasses a variety of glycemic abnormalities that are commonly referred to as 'prediabetes'. While intensive lifestyle interventions are the cornerstone of T2D prevention, developing safe, cost-effective adjunct therapeutic strategies is a clinically relevant goal. Cinnamon supplementation has been shown to improve fasting plasma glucose in patients with T2D. This placebo-controlled, randomized study will determine if cinnamon improves glucose homeostasis in patients with prediabetes over a 12-week period.

DETAILED DESCRIPTION:
BACKGROUND: The transition from normal glucose tolerance and insulin sensitivity to overt type 2 diabetes (T2D) encompasses a variety of glycemic abnormalities that are commonly referred to as 'prediabetes'. In 2003, 314 million people (8.2% of the adult population) had prediabetes, and this number is projected to increase to 472 million (9.0% of the adult population) by 2025. Approximately 40-50% of individuals with prediabetes have been reported to develop T2D within 10 years.

While intensive lifestyle interventions remain the cornerstone of T2D prevention, targeted pharmacotherapy has been shown to be effective and may be considered in high-risk patients. Several antidiabetic medications prevent or, at least, delay the progression from prediabetes to diabetes, including metformin, α-glucosidase inhibitors or pioglitazone. However, cost, potential adverse effects, and secondary failure in the long-term have often limited the widespread use of these and other newer antidiabetic drugs in patients with prediabetes. For instance 10 to 20% of metformin-treated patients experience gastrointestinal side effects (nausea, vomiting, and diarrhea) leading to its discontinuation, whereas the use pioglitazone is often complicated by weight gain and increased risk of fractures.

In this context, efficacious, cost-effective, and safe adjunct therapeutics for T2D prevention are highly desirable. The present trial proposes to test the effects of cinnamon in patients with prediabetes.

RATIONALE: Several randomized controlled studies have addressed the effects of cinnamon on changes in glycated hemoglobin (HbA1c) and fasting plasma glucose (FPG) in adult patients with T2D. Almost all studies showed a significant 10-20% decrease in FPG from baseline and improvements in HbA1c, although the latter change often did not achieve statistical significance. These findings in patients with T2D provide the rational to test whether cinnamon exerts similar beneficial effects in patients with prediabetes.

STUDY DESIGN: This is a multi-center placebo-controlled, randomized (1:1), double masked trail to assess the effects of cinnamon (cinnamomum burmannii) on glucose homeostasis over a 12- week period. FPG, HbA1c, and other measures of glucose metabolism will be collected at baseline, after 6 weeks, and at the end of the 12-week study period. Participants will be prompted to report Adverse Events (AE) at the study visits or anytime during the study period.

OUTCOMES: The primary outcome for the Cinnamon Trial is a change in the FPG level from baseline to week 12 of treatment, as compared to placebo. Secondary outcomes include change in the FPG from baseline to week 6 of treatment, and change from baseline in plasma glucose at 2 hours and area under the curve-glucose during a 75-gram oral glucose tolerance test to week 12. Data will be analyzed using the "intent-to-treat" approach, which includes all randomized subjects with at least one post-baseline FPG measurement; the supplementation group assignment will not be altered based on the subject's adherence to the regimen.

SAMPLE SIZE DETERMINATION: Anticipating an absolute change in FPG smaller than what observed in previous studies in patients with T2D, 10 patients with prediabetes in total entering a two-treatment parallel-design study will provide 90% probability of detecting a true between-treatment difference in FPG means of 22 mg/dl with standard deviation of 10 mg/dl, using a paired two-sided comparison with type 1 error of 0.05. To allow for up to 20% dropout, 12 patients in total will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 20 - 70 years old at screening
2. Meet at least one of the following criteria of Prediabetes according to the 2016 American Diabetes Association criteria:

   1. Impaired Fasting Glucose (IFG [100-125 mg/dL])
   2. Impaired Glucose Tolerance (IGT [2-h plasma glucose: 140-199 mg/dL based on 75-g OGTT])
   3. HbA1c between 5.7-6.4%
3. Willingness to provide informed consent and follow all study procedures, including attending all scheduled visits.

Exclusion Criteria:

1. Documented diabetes mellitus diagnosed by a physician and confirmed by other clinical data.
2. Previous use of any antidiabetic medication.
3. Cardiovascular disease within 6 months of the study commencement including arrhythmia, congestive heart failure, myocardial infarction or pacemaker placement.
4. History of uncontrolled hypertension (defined as systolic blood pressure > 150 mmHg or diastolic blood pressure > 95 mmHg on three or more assessments on more than 1 day). If the patient is on blood pressure medications, dosing should be stable for at least 4 weeks prior to randomization.
5. Cancer diagnosis requiring treatment in the past 5 years
6. Chronic kidney disease stage 3-5 (estimated glomerular filtration rate < 60; based on MDRD formula or creatinine ≥ 1.4 for men or >1.3 mg/dL for women, or a urine protein ≥ 2+)
7. Known liver disease or elevation of AST, ALT, or GGT > 2.50 × upper limit of normal at screening.
8. Other gastrointestinal diseases (including pancreatitis and inflammatory bowel disease)
9. Participation in other clinical trials within 2 months.
10. Surgery within 30 days prior to screening.
11. Pulmonary disease with dependence on oxygen or daily use of bronchodilators.
12. Chronic infections (e.g., human immune-deficiency virus (HIV) or active tuberculosis)
13. Allergy or hypersensitivity to any of the ingredients in the test products.
14. Cognitive impairment or any other reason to expect the patient would have difficulty complying with study protocol
15. Excessive alcohol intake defined as greater than 3 units of alcohol per day.
16. Use of weight loss drugs (e.g., lorcaserin [Belviq]; phentermine/topiramate [Qsymia], liraglutide [Saxenda], Xenical [orlistat], Meridia [sibutramine], Acutrim [phenylpropanol-amine], or similar over-the-counter medications) within 3 months of the screening visit.
17. Intentional weight loss of ≥ 10 lbs in the previous 6 months.
18. Use of dietary supplements that may have glucose-lowering effects (e.g. Sesame, Polygonatum odoratum, Chromium, Vanadium).
19. Concurrent enrollment in a weight loss program, such as Weight Watchers.
20. Other endocrine disorders affecting glucose metabolism including Cushing' syndrome, acromegaly, hyperthyroidism, hypothyroidism or adrenal insufficiency.
21. Fasting plasma triglyceride >500 mg/dl.
22. Oral corticosteroids within 3 months.
23. Pregnancy and/ or Lactation: Women of childbearing potential will be required to have a negative urine pregnancy test and to use contraception measures during the study and for at least 1 month after participating in the study. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
24. Moderate anemia, defined as hemoglobin <10.9 in both men and women based on WHO criteria

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose at 12 weeks | 12 weeks
  Change from baseline in fasting plasma glucose at 12 weeks

SECONDARY OUTCOMES:
Fasting plasma glucose at 6 weeks | 6 weeks
  Change from baseline in fasting plasma glucose at 6 weeks
2-hour plasma glucose during OGTT (oral glucose tolerance test) | 12 weeks
  Change from baseline in plasma glucose obtained 2 hours during OGTT at 12 weeks
Area under the curve-glucose during OGTT (oral glucose tolerance test) | 12 weeks
  Change from baseline in area under the curve of plasma glucose during OGTT at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giulio R Romeo, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Medagama AB. The glycaemic outcomes of Cinnamon, a review of the experimental evidence and clinical trials. Nutr J. 2015 Oct 16;14:108. doi: 10.1186/s12937-015-0098-9. PMID 26475130
- [Background] Hlebowicz J, Hlebowicz A, Lindstedt S, Bjorgell O, Hoglund P, Holst JJ, Darwiche G, Almer LO. Effects of 1 and 3 g cinnamon on gastric emptying, satiety, and postprandial blood glucose, insulin, glucose-dependent insulinotropic polypeptide, glucagon-like peptide 1, and ghrelin concentrations in healthy subjects. Am J Clin Nutr. 2009 Mar;89(3):815-21. doi: 10.3945/ajcn.2008.26807. Epub 2009 Jan 21. PMID 19158209
- [Background] Khan A, Safdar M, Ali Khan MM, Khattak KN, Anderson RA. Cinnamon improves glucose and lipids of people with type 2 diabetes. Diabetes Care. 2003 Dec;26(12):3215-8. doi: 10.2337/diacare.26.12.3215. PMID 14633804